CLINICAL TRIAL: NCT02733354
Title: Impact of Lifestyle Scenario Demonstration on Patients'Decision-making of Dialysis Modality
Brief Title: Lifestyle Scenario Demonstration on Dialysis Modality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Xuanyi Du, chief physician, The Second Affiliated Hospital of Harbin Medical University
Other Study IDs: 2ndHarbinMU
Record Dates: First submitted 2016-04-06; First posted 2016-04-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Dialysis Mode Life Scenarios

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control Group: Control Group:perform routine oral education.Both groups were asked to complete kidney disease knowledge questionnaire before education.
- Intervention Group: Intervention Group ：On the basis of Control Group, watching video demonstration of each type of dialysis. The videos were based on real cases, showing patients with peritoneal and hemodialysis life modes, lasting for 20 minutes respectively for each type of dialysis. Both groups were asked to complete kidney disease knowledge questionnaire before education.
  Interventions: Device: watch viedo

INTERVENTIONS:
Device: watch viedo
  Groups: Intervention Group

SUMMARY:
Based on real cases, daily life scenarios of peritoneal dialysis and hemodialysis patients were shooted and edited into video films, including environment of home dialysis, dietary patterns, water intake, sports mode, daily work, short time of travel and other activities, covering a certain natural day of either peritoneal or hemodialysis and some important time points in the way of life, such as nursing and treatment for common complications of the corresponding dialysis mode. The videos will also show the advantages and disadvantages of the two modes of dialysis. According to their actual living conditions, patients will decide the right dialysis modality that suite them well, thus improving dialysis compliance and psychological adaptability.

DETAILED DESCRIPTION:
Based on real cases, daily life scenarios of peritoneal dialysis and hemodialysis patients were shooted and edited into video films, including environment of home dialysis, dietary patterns, water intake, sports mode, daily work, short time of travel and other activities, covering a certain natural day of either peritoneal or hemodialysis and some important time points in the way of life, such as nursing and treatment for common complications of the corresponding dialysis mode. The videos will also show the advantages and disadvantages of the two modes of dialysis. According to their actual living conditions, patients will decide the right dialysis modality that suite them well, thus improving dialysis compliance and psychological adaptability.

By "informed decision score" questionnaire, comparison of two groups of patients on dialysis awareness of the pattern and ratio of patients choosing hemodialysis and peritoneal dialysis were performed. Dialysis mode conversion rates of the two groups were finally calculated and the correlation between awareness of dialysis modality and conversion rates of dialysis methods was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* CKD（chronic kidney disease） stage 5 patients with replacement therapy indications, age≥ 18 years, ≤70 years
* without any contraindications of peritoneal dialysis or hemodialysis

Exclusion Criteria:

* Age> 70 years or <18 years old
* contraindications of peritoneal dialysis or hemodialysis
* Patients who cannot be followed well after dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD 5 patients,prepare for dialysis, aged between 18 to 70 years old, male or female,
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Conversion rates | two years

SECONDARY OUTCOMES:
Informed Decision Score | two years